CLINICAL TRIAL: NCT03084692
Title: Feasibility and Preliminary Efficacy of a Combined Therapeutic Yoga and Resistance Exercise Intervention for Individuals With Lung Cancer and Their Caregivers
Brief Title: Therapeutic Yoga and Resistance Exercise for Lung Cancer
Acronym: ASSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-17-0049
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer
Keywords: caregiver; lung cancer; yoga; resistance exercise
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: A single group before and after intervention study design will be used for this pilot feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Yoga and Resistance Exercise (Experimental): The individuals with lung cancer and their caregivers will participate in a combined intervention of yoga and resistance exercise for 8-week, two times/week. The dyad will attend a one-hour resistance exercise intervention at the start of the week and a one-hour yoga class with a break of one day between both interventions. The resistance exercise training will involve one-on-one personal exercise session, while the yoga intervention will be offered in a class setting. The participants will be allowed to make up for any missed resistance exercise session based on the available time. Pamphlets will be given demonstrating breathing exercises, meditation, postures, and core resistance exercises to facilitate programming.
  Interventions: Behavioral: Therapeutic Yoga and Resistance Exercise

INTERVENTIONS:
Behavioral: Therapeutic Yoga and Resistance Exercise — Combined Program of Yoga and Resistance Exercise

SUMMARY:
The purpose of the study is to determine the feasibility and preliminary efficacy of a combined therapeutic yoga and resistance exercise intervention for individuals with lung cancer and their caregivers. The investigators aim is to help reduce the fear of exercise by tailoring the program to meet the specific needs of the survivor with lung cancer. The investigators want to see whether individuals with lung cancer and their caregivers are interested in participating in this type of program, and if they are able to attend the intervention sessions and complete the program. The investigators also plan to study the preliminary effects of therapeutic yoga and resistance exercise on fitness outcomes for both individuals with lung cancer and their caregivers.

DETAILED DESCRIPTION:
To determine the feasibility of a combined therapeutic yoga and resistance exercise intervention for lung cancer survivors and their caregivers. A single group before and after intervention study design will be used for this pilot feasibility trial. Brochures and information about the study will be distributed at the Cross Cancer Institute, and interested individuals will be screened for eligibility. A convenient sampling technique will be used to recruit individuals with lung cancer and their caregiver. Participants deemed eligible to take part in the study will provide written informed consent to participate in the study and will undergo baseline testing. The intervention will be carried out over a period of 8 weeks. The feasibility outcomes will include eligibility rate, completion rate, adherence rate and adverse events. Dyspnea will be the primary self-reported outcome to be measured for individuals with lung cancer. The secondary outcomes will include fatigue, shoulder range of motion, chest expansion, and muscular strength. The outcome measures for the caregivers will include quality of life (QoL) and muscular strength.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Primary Lung Cancer Stage I-IV (all stages)
2. Any form of Lung cancer included: Small Cell Lung Cancer and Non-Small Cell Lung Cancer
3. Age: 18 years or above
4. Patients at any time point during treatment: ongoing treatment, completed treatment or recently diagnosed and about to start treatment
5. Karnofsky Performance Status ≥ 50 (Appendix A)
6. Life expectancy at least one year -

Exclusion Criteria:

1. Metastatic lung disease that would preclude safe exercise prescription
2. Secondary Lung cancer due to metastasis from other parts of body
3. Co-morbid conditions such as diabetes, congestive heart failure, dementia, cerebrovascular diseases.
4. Individuals who would be unsafe to participate in an intervention program.
5. Unable to provide consent in English
6. Unable to complete either testing or intervention components (e.g. extended holiday)

Caregiver eligibility: Caregivers will be screened using the PAR-Q + questionnaire and will be required to obtain approval from a family physician should any safety concerns be identified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Completion Rate | Up to 24 weeks
  Completion rate is defined as the number of participants successfully completing the baseline assessment, intervention, and the post-intervention assessment.

SECONDARY OUTCOMES:
Dyspnoea Visual Analogue Scale | 8 weeks
  Visual Analogue Scale used to measure subjective breathlessness of a horizontal 10-cm line with phrases at both ends of the scale demonstrating minimum and maximum level of breathlessness.
Dyspnoea-12 | 8 weeks
  The dyspnea-12 consists of 12 item scale to which patients respond about their general perception of their current state. It quantifies breathlessness using descriptions by patients of both physical and affective aspects of dyspnoea.
Functional Assessment of Cancer Therapy: Fatigue Scale (FACT-F) | 8 weeks
  The FACT-F was developed to measure fatigue in oncology patients with anemia. It has 13 items, which cover physical fatigue, functional fatigue, emotional fatigue, and social consequences of fatigue.
Chest expansion (centimetres) | 8 weeks
  The circumference of the chest is measured after an inspiration and an expiration using a tape at the level xiphisternum in standing position, using two different arm positions: hands on head and arms at the side.
Shoulder Range of Motion (degrees) | 8 weeks
  Active Flexion and Abduction will be measured using a handheld goniometer with the participant in a sitting position.
Muscular strength | 8 weeks
  All participants, the individuals with lung cancer and their caregivers will perform a 1RM test before and after the 8-week intervention, to measure the changes in their muscle strength of upper extremity and lower extremity on a bench press, seated row, and a leg press.
Pulmonary Function Testing | 8 weeks
  The lung volumes and capacities will be measured using the spirometer in a sitting position. The forced expiratory volume in one second (fev1) and the forced vital capacity (fvc) will be measured.
CareGiver Oncology Quality of Life (CarGOQoL) questionnaire (Caregivers only) | 8 weeks
  The CareGiver Oncology Quality of Life (CarGOQoL) questionnaire is a 29-item, multidimensional, self-administered questionnaire.
Chalder Fatigue Scale (Caregivers only) | 8 weeks
  Chalder Fatigue Scale is an 11 item scale to assess symptoms of fatigue such as tiredness, sleepiness, lack of energy, lack of strength in the muscles, difficulties in concentration and memory.
Adherence Rate | up to 8 weeks
  Attendance at exercise sessions
Recruitment rate | 24 weeks
  The number of participants agreeing to participate divided by the total number eligible
Adverse Event | up to 24 weeks
  Incidence of serious and non-serious adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNeely, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time.